CLINICAL TRIAL: NCT03949413
Title: Correlation Between Balance and Attention in Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Lecturer in Department of Physical Therapy for Pediatric Disorders, Faculty of Physical Therapy, Delta University for Science and Technology
Other Study IDs: DeltaUPT1
Record Dates: First submitted 2019-05-08; First posted 2019-05-14 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Attention Deficit Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group (A): 30 normal children
- study Group (B): 30 children from both sexes (22 boys and 8 girls) with attention deficit hyperactivity disorder (ADHD)

SUMMARY:
Objective: The purpose of the current study was to investigate balance in children with attention deficit hyperactivity disorder compared to normal subjects. Furthermore, it studied the relationship between their balance and the total percentile scores of the ADHD Rating Scale IV.

DETAILED DESCRIPTION:
Objective: The purpose of the current study was to investigate balance in children with attention deficit hyperactivity disorder contrasted to normal subjects. Furthermore, it studied the relationship between their balance and the total percentile scores of ADHD Rating Scale-IV.

Design: The study was a cross-sectional design. Methods: Sixty children were involved in this research from both sexes (42 boys and 18 girls) with age ranged from 60 to 84 months. They were subdivided into two groups based on the ADHD Rating Scale-IV. The control group included 30 normally developed children from both sexes (20 boys and 10 girls) with a mean age of 67.53 ± 1.41 months, and the total percentile scores of ADHD Rating Scale-IV ≤ 50. The study group comprised of 30 children from both sexes (22 boys and 8 girls) with attention deficit hyperactivity disorder (ADHD) with a mean age of 68.60 ± 4.62 months. The total percentile scores of ADHD Rating ScaleIV were ≥ 93. Both groups were investigated for their balance by Pediatric Balance Scale (PBS).

ELIGIBILITY:
Sixty children were involved in the present research from both sexes (42 boys and 18 girls) which were subdivided into two equal groups (control and study groups). They were recruited from different kindergartens at Cairo, Egypt, based on the following criteria:

inclusive criteria:

* age ranged from 60 to 84 months.
* selected from both sex.
* Children in the study group with attention deficit hyperactivity disorder (ADHD) based on the ADHD Rating Scale-I with total percentile scores ≥ 93, Children in control group normally developed with total percentile scores of ADHD Rating Scale-IV ≤ 50.

exclusive criteria:

- no history of cerebral palsy, epilepsy or head trauma.

Ages: 60 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sixty children were involved in the present research from both sexes (42 boys and 18 girls) with age ranged from 60 to 84 months, which were subdivided into two groups (control and study groups). They were recruited from different kindergartens at Cairo, Egypt
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale-IV checklist, school version | At the baseline evaluation.
  Both groups were investigated by the ADHD Rating Scale-IV checklist, school version to know if the child was diagnosed with ADHD or rule out.
Pediatric Balance Scale (PBS) | At the baseline evaluation.
  Both groups were assessed for their balance by PBS

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Kindergartens, Cairo
  - Amira Hussin Mohammed, Gamasa